CLINICAL TRIAL: NCT02926664
Title: Prognostic Value of Quick Sequential Organ Failure Assessment Kinetics After Fluids Challenge in the Emergency Department
Brief Title: Delta qSOFA for Risk Stratification in Emergency Infected Patients
Acronym: DELTASCREEN
Status: Completed | Type: Observational
Sponsor: Societe Française de Medecine d'urgence (Other)
Responsible Party: Principal Investigator, Yonathan Freund, Associate professor, Societe Française de Medecine d'urgence
Other Study IDs: DeltaSCREEN
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: measurement of qSOFA — qSOFA will be measured at H0, H1 and H3

SUMMARY:
The study will investigate the prognostic value of qSOFA (quick Sequential Organ Failure Assessment) kinetics between H0 and H1, and between H0 and H3 in patients with suspicion of Sepsis, i.e. an initial qSOFA of at least of 2.

DETAILED DESCRIPTION:
qSOFA has been reported as a good tool for risk stratification in the ED for patients with infection.

However, it is not clear whether qSOFA remains stable during the ED stay, nor whether its kinetics can have prognostic added value.

Patients with a qSOFA of at least 2 in the ED, and suspicion of infection will be included.

After treatment is initiated and fluids challenge performed, we will collect qSOFA value at 1 hour and 3 hours.

Our hypothesis is that a decrease in qSOFA between H0 and H3 is associated with better outcome. We assume that 50% of patients will have a deltaqSOFA >0, with an overall mortality of 23% (according to previous cohort). Under the hypothesis of difference of at least 15% in mortality between the two groups (DeltaqSOFA > 0 and Delta qSOFA<=0), with a power of 90% and an alpha of 0.05, we need to recruit 322 patients.

ELIGIBILITY:
Inclusion Criteria:

* suspicion of infection by the emergency physicians
* at least two of the following criteria : respiratory rate <= 22, systolic blood pressure <= 100 mmHg and altered mental status

Exclusion Criteria:

* Infection ruled out by the expert after chart review
* patient who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients in the ED who presents with suspicion of infection AND a qSOFA of at least 2.
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2016-10; Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 60 days

SECONDARY OUTCOMES:
ICU admission more than 72 hours | 60 days
ICU admission | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan Freund, Principal Investigator — Emergency Department - hopital pitie salpetriere, Paris, France
Locations (10):
- Cliniques St Luc, Brussels, Belgium
- France (8):
  - CHU Nimes, Nîmes
  - Cochin, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Pitié-Salpêtrière, Paris
  - Hopital Tenon, Paris
  - Lariboisière, Paris
  - Saint Antoine, Paris
  - CHU Strasbourg, Strasbourg
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
data will be available upon request to the principal investigator